CLINICAL TRIAL: NCT02611323
Title: A Phase Ib/II Study Evaluating the Safety and Efficacy of Obinutuzumab in Combination With Polatuzumab Vedotin and Venetoclax in Patients With Relapsed or Refractory Follicular Lymphoma and Rituximab in Combination With Polatuzumab Vedotin and Venetoclax in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Obinutuzumab, Rituximab, Polatuzumab Vedotin, and Venetoclax in Relapsed or Refractory Follicular Lymphoma (FL) or Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29833; 2015-001998-40 (EudraCT Number)
Record Dates: First submitted 2015-11-19; First posted 2015-11-20 (Estimated); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — obinutuzumab; Rituximab; polatuzumab vedotin; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose-Escalation Cohort: FL (Experimental): Participants with relapsed or refractory FL will receive 18 weeks of induction treatment with polatuzumab vedotin and venetoclax at escalating doses to identify the recommended Phase 2 dose (RP2D) for polatuzumab vedotin and venetoclax when combined with a fixed dose of obinutuzumab. Those who achieve CR, PR, or SD at the EOI will be eligible to receive a 24-month maintenance regimen consisting of 8 months of venetoclax and 24 months of obinutuzumab.
  Interventions: Drug: Obinutuzumab; Drug: Polatuzumab Vedotin; Drug: Venetoclax
- Dose-Escalation Cohort: DLBCL (Experimental): Participants with relapsed or refractory DLBCL will receive 18 weeks of induction treatment. Venetoclax will be administered at escalating doses to identify the RP2D of venetoclax when combined with fixed doses of polatuzumab vedotin and rituximab. Those who achieve CR or PR at the EOI will be eligible to receive an 8-month consolidation regimen consisting of venetoclax and rituximab.
  Interventions: Drug: Rituximab; Drug: Polatuzumab Vedotin; Drug: Venetoclax
- Expansion Cohort: FL (Experimental): Participants with relapsed or refractory FL will receive 18 weeks of induction treatment with polatuzumab vedotin and venetoclax at the RP2D identified during the dose-escalation phase, in addition to obinutuzumab. Those who achieve CR, PR, or SD at the EOI will be eligible to receive a 24-month maintenance regimen consisting of 8 months of venetoclax and 24 months of obinutuzumab.
  Interventions: Drug: Obinutuzumab; Drug: Polatuzumab Vedotin; Drug: Venetoclax
- Expansion Cohort: DLBCL (Experimental): Participants with relapsed or refractory DLBCL will receive 18 weeks of induction treatment. Venetoclax will be administered at the RP2D identified during the dose-escalation phase, in addition to polatuzumab vedotin and rituximab. Those who achieve CR or PR at the EOI will be eligible to receive an 8-month consolidation regimen consisting of venetoclax and rituximab.
  Interventions: Drug: Rituximab; Drug: Polatuzumab Vedotin; Drug: Venetoclax

INTERVENTIONS:
Drug: Obinutuzumab — Participants will receive a fixed dose of obinutuzumab, 1000 milligrams (mg) via intravenous (IV) infusion to be given on Days 1, 8 and 15 of Cycle 1 and on Day 1 of Cycles 2 to 6. Cycle length will be 21 days. For eligible participants, post-induction treatment may be given at a dose of 1000 mg via IV infusion on Day 1 of every other month (starting from Month 2) for up to 24 months, until disease progression or unacceptable toxicity.
  Arms: Dose-Escalation Cohort: FL; Expansion Cohort: FL
Drug: Rituximab — Participants will receive a fixed dose of rituximab, 375 milligrams per square meter (mg/m^2) via IV infusion to be given on Day 1 of Cycles 1 to 6. Cycle length will be 21 days. For eligible participants, post-induction treatment may be given at a dose of 375 mg/m^2 via IV infusion on Day 1 of every other month (starting from Month 2) for up to 8 months, until disease progression or unacceptable toxicity.
  Arms: Dose-Escalation Cohort: DLBCL; Expansion Cohort: DLBCL
Drug: Polatuzumab Vedotin — Participants will receive polatuzumab vedotin via IV infusion at doses of 1.4 or 1.8 milligrams per kilogram (mg/kg) (for FL), and 1.8 mg/kg (for DLBCL) on Day 1 of each 21-day cycle for up to 18 weeks during induction treatment. Polatuzumab vedotin will not be given during the post-induction period.
Drug: Venetoclax — Participants will receive venetoclax film-coated tablets at doses of 200, 400, 600, or 800 mg (for FL), and 400, 600, or 800 mg (for DLBCL) on Days 1 to 21 of each 21-day cycle. Post-induction venetoclax may continue for up to 8 months, until disease progression or unacceptable toxicity.

SUMMARY:
This study will evaluate the safety, efficacy, and pharmacokinetics of induction treatment with obinutuzumab, polatuzumab vedotin, and venetoclax in participants with relapsed or refractory FL, and with rituximab, polatuzumab vedotin, and venetoclax in participants with DLBCL. Participants with FL who achieve complete response (CR), partial response (PR), or stable disease (SD) at the end of induction therapy will receive post-induction treatment with obinutuzumab and venetoclax, and participants with DLBCL who achieve CR or PR at the end of induction (EOI) will receive post-induction treatment with rituximab and venetoclax.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* For obinutuzumab + polatuzumab vedotin + venetoclax treatment group, relapsed or refractory FL after treatment with at least one prior chemoimmunotherapy regimen that included an anti-cluster of differentiation 20 (CD20) (anti-CD20) monoclonal antibody (mAb) and for which no other more appropriate treatment option exists, as determined by the investigator
* For rituximab + polatuzumab vedotin + venetoclax treatment group, relapsed or refractory DLBCL after treatment with at least one prior chemoimmunotherapy regimen that included an anti-CD20 mAb and for which no curative option exists as determined by the investigator
* At least one bidimensionally measurable lesion

Exclusion Criteria:

* Known CD20-negative status at relapse or progression
* Prior allogeneic stem cell transplantation (SCT), or autologous SCT within 100 days prior to Day 1 of Cycle 1
* Grade 3b FL
* History of transformation of indolent disease to DLBCL
* Current use of systemic corticosteroids greater than (>) 20 mg prednisone per day (or equivalent); or prior anti-cancer therapy to include: radioimmunoconjugate within 12 weeks; mAb or antibody-drug conjugate within 4 weeks; or radiotherapy/chemotherapy/hormone therapy/targeted small-molecule therapy within 2 weeks prior to Day 1 of Cycle 1
* Central nervous system (CNS) disease
* Active infection
* Actual or potential cytochrome P450 (CYP) 3A interactions including: requirement for warfarin; use of strong and moderate CYP3A inhibitors or inducers within 7 days prior to first dose of venetoclax; or consumption of grapefruit, Seville oranges, or star fruit within 3 days prior to first dose of venetoclax
* Positive for human immunodeficiency virus (HIV) or hepatitis B or C
* Receipt of a live virus vaccine within 28 days prior to Day 1 of Cycle 1
* Poor hematologic, renal, or hepatic function
* Pregnant or lactating women
* Life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (10):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - Memorial Healthcare System, Pembroke, Florida
  - Emory Univ Winship Cancer Inst, Atlanta, Georgia
  - University of Louisville Hospital; The James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Inst., Buffalo, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Scott and White, Temple, Texas
- Australia (6):
  - Royal North Shore Hospital; Haematology Department, St Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peter MacCallum Cancer Center, North Melbourne, Victoria
- Italy (7):
  - Papa Giovanni Hospital XXIII, Bergamo, Emilia-Romagna
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola, Emilia-Romagna
  - UO Ematologia, Ospedale S.Maria delle Croci, Ravenna, Emilia-Romagna
  - Ospedale Infermi U.O. Ematologia, Rimini, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - SCDU Ematologia, Novara, Piedmont
  - A.O.U. Citta' Della Salute E Della Scienza-P.O. Molinette;S.C. Ematologia, Turin, Piedmont

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 23 investigative centers in Australia, Italy, and the United States from 09 March 2016 up to 04 August 2022. The study consisted of two phases: a dose-escalation phase and a dose-expansion phase. All eligible participants in both dose-escalation and expansion phases received induction treatment, and post-induction treatment as indicated.
Pre-assignment Details: A total of 133 participants with relapsed or refractory (R/R) follicular lymphoma (FL) and R/R diffuse large B-cell lymphoma (DLBCL) were enrolled in this study. Out of the 133, two participants did not receive any study treatment. Of the 131 treated participants, 74 participants with FL received Obinutuzumab (G) in combination with polatuzumab vedotin (P) and venetoclax (V) and 57 participants with DLBCL received rituximab (R) in combination with polatuzumab vedotin and venetoclax.
Groups:
- FL Dose Escalation: 1.4P+400V+1000G: Participants received venetoclax, 400 milligrams (mg), orally, once daily (QD) on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with obinutuzumab, 1000 mg, intravenous (IV) infusion, on Days 1, 8 and 15 of Cycle 1 and thereafter on Day 1 of Cycles 2-6 and polatuzumab vedotin, 1.4 milligrams per kilograms (mg/kg), IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved complete response (CR), partial response (PR), or stable disease (SD) at end of induction (EOI) received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received venetoclax, 400 mg, QD, for up to 8 months and obinutuzumab, 1000 mg on Day 1 of every other month (1 month=28 days) starting from Month 2 for up to 24 months.
- FL Dose Escalation: 1.4P+200V+1000G: Participants received venetoclax, 200 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with obinutuzumab, 1000 mg, IV infusion, on Days 1, 8 and 15 of Cycle 1 and thereafter on Day 1 of Cycles 2-6 and polatuzumab vedotin, 1.4 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received venetoclax, 200 mg, QD, for up to 8 months and obinutuzumab, 1000 mg on Day 1 of every other month (1 month=28 days) starting from Month 2 for up to 24 months.
- FL Dose Escalation: 1.8P+400V+1000G: Participants received venetoclax, 400 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with obinutuzumab, 1000 mg, IV infusion, on Days 1, 8 and 15 of Cycle 1 and thereafter on Day 1 of Cycles 2-6 and polatuzumab vedotin, 1.8 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received venetoclax, 400 mg, QD, for up to 8 months and obinutuzumab, 1000 mg on Day 1 of every other month (1 month=28 days) starting from Month 2 for up to 24 months.
- FL Dose Escalation: 1.4P+600V+1000G: Participants received venetoclax, 600 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with obinutuzumab, 1000 mg, IV infusion, on Days 1, 8 and 15 of Cycle 1 and thereafter on Day 1 of Cycles 2-6 and polatuzumab vedotin, 1.4 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received venetoclax, 600 mg, QD, for up to 8 months and obinutuzumab, 1000 mg on Day 1 of every other month (1 month=28 days) starting from Month 2 for up to 24 months.
- FL Dose Escalation: 1.8P+600V+1000G: Participants received venetoclax, 600 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with obinutuzumab, 1000 mg, IV infusion, on Days 1, 8 and 15 of Cycle 1 and thereafter on Day 1 of Cycles 2-6 and polatuzumab vedotin, 1.8 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received venetoclax, 600 mg, QD, for up to 8 months and obinutuzumab, 1000 mg on Day 1 of every other month (1 month=28 days) starting from Month 2 for up to 24 months.
- FL Dose Escalation: 1.8P+800V+1000G; FL: Dose Expansion: 1.8P+800V+1000G: Participants received venetoclax, 800 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with obinutuzumab, 1000 mg, IV infusion, on Days 1, 8 and 15 of Cycle 1 and thereafter on Day 1 of Cycles 2-6 and polatuzumab vedotin, 1.8 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received venetoclax, 800 mg, QD, for up to 8 months and obinutuzumab, 1000 mg on Day 1 of every other month (1 month=28 days) starting from Month 2 for up to 24 months.
- DLBCL: Dose Escalation: 1.8P+400V+375R: Participants received venetoclax, 400 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with rituximab, 375 milligrams per square meter (mg/m^2), IV infusion, on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR or PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 8 months. During consolidation treatment participants received venetoclax, 400 mg, QD, for up to 8 months and rituximab, 375 mg/m^2 on Day 1 of every other month (1 month=28 days) starting from Month 2 up to 8 months.
- DLBCL Dose Escalation: 1.8P+600V+375R: Participants received venetoclax, 600 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with rituximab, 375 mg/m^2, IV infusion, on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR or PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 8 months. During consolidation treatment participants received venetoclax, 600 mg, QD, for up to 8 months and rituximab, 375 mg/m^2 on Day 1 of every other month (1 month=28 days) starting from Month 2 up to 8 months.
- DLBCL Dose Escalation: 1.8P+800V+375R; DLBCL Dose Expansion: 1.8P+800V+375R: Participants received venetoclax, 800 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with rituximab, 375 mg/m^2, IV infusion, on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR or PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 8 months. During consolidation treatment participants received venetoclax, 800 mg, QD, for up to 8 months and rituximab, 375 mg/m^2 on Day 1 of every other month (1 month=28 days) starting from Month 2 up to 8 months.
Period: Overall Study
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Started | 7 | 3 | 3 | 3 | 9 | 8 | 41 | 3 | 6 | 8 | 40
Completed | 2 | 2 | 3 | 3 | 8 | 7 | 30 | 2 | 2 | 0 | 11
Not Completed | 5 | 1 | 0 | 0 | 1 | 1 | 11 | 1 | 4 | 8 | 29
Not completed — Death | 3 | 1 | 0 | 0 | 1 | 1 | 8 | 0 | 4 | 6 | 26
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2
Not completed — Found Another Malignancy After Starting Trial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety-evaluable population included all participants who received at least one dose of any component of the combination.
Groups:
- FL Dose Escalation: 1.4P+400V+1000G: Participants received venetoclax, 400 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with obinutuzumab, 1000 mg, IV infusion, on Days 1, 8 and 15 of Cycle 1 and thereafter on Day 1 of Cycles 2-6 and polatuzumab vedotin, 1.4 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received venetoclax, 400 mg, QD, for up to 8 months and obinutuzumab, 1000 mg on Day 1 of every other month (1 month=28 days) starting from Month 2 for up to 24 months.
- Total: Total of all reporting groups
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R | Total
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 41 | 3 | 6 | 8 | 40 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (6.8) | 61.3 (8.5) | 56.7 (13.6) | 58.3 (10.3) | 64.6 (6.1) | 58.0 (11.9) | 62.2 (11.3) | 56.0 (16.5) | 58.7 (17.4) | 67.4 (15.2) | 65.8 (9.6) | 62.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 0 | 4 | 4 | 20 | 2 | 4 | 5 | 18 | 61
  Male | 4 | 2 | 3 | 3 | 5 | 4 | 21 | 1 | 2 | 3 | 22 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 4
  White | 7 | 3 | 3 | 3 | 8 | 7 | 34 | 2 | 6 | 6 | 30 | 109
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 6 | 0 | 0 | 1 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 7 | 3 | 3 | 3 | 8 | 8 | 30 | 3 | 6 | 7 | 31 | 109
  Not Stated | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 0 | 0 | 1 | 6 | 14
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With CR at EOI Determined by an Independent Review Committee (IRC) on the Basis of Positron Emission Tomography (PET) and Computed Tomography (CT) Scans
Description: CR at EOI was assessed by the IRC according to modified Lugano Response Criteria (MLRC) for Malignant Lymphoma 2014 using PET-CT scan. Per MLRC, CR was defined as complete metabolic response (MR) in lymph nodes and extra lymphatic sites (ELS) with a score of 1, 2, or 3, with or without a residual mass on PET 5-point scale (5-PS), where 1=no uptake above background; 2= uptake ≤mediastinum; 3= uptake > mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions. No new lesions; no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. 90% confidence interval (CI) for percentage of responders was calculated using Clopper-Pearson method. Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 23 weeks) (1 cycle=21 days)
Population: Efficacy evaluable population included participants in the dose expansion arms who received at least one dose of any component of the combination. As pre-specified in the protocol, participants who received polatuzumab vedotin and venetoclax at recommended phase 2 dose (RP2D) in dose-escalation phase were also analyzed in addition to expansion phase participants for efficacy analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 8 | 41 | 8 | 40
percentage of participants | 100 [68.77 to 100.00] | 51.2 [37.44 to 64.86] | 25 [4.64 to 59.97] | 32.5 [20.41 to 46.63]

2. Primary Outcome: FL Cohorts: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any new disease or worsening of an existing disease were also considered as AEs. An SAE was defined as any AE that was fatal, life threatening, requires prolonged inpatient hospitalization, resulted in significant disability or resulted in a congenital anomaly to a mother exposed to study treatment. AEs and SAEs were reported based on the National Cancer Institute Common Terminology Criteria for AEs, version 4.0 (NCI-CTCAE, v4.0). Percentages have been rounded off to the first decimal point.
Time Frame: From study start to 24 months after last dose of study drug (approximately 56 months)
Population: Safety-evaluable population included all participants who received at least one dose of any component of the combination. The safety-evaluable population in the FL cohorts were assessed in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 41
percentage of participants
  AEs | 100 | 100 | 100 | 100 | 100 | 100 | 100
  SAEs | 57.1 | 33.3 | 33.3 | 0 | 22.2 | 75.0 | 34.1

3. Primary Outcome: DLBCL Cohorts: Percentage of Participants With AEs and SAEs
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any new disease or worsening of an existing disease were also considered as AEs. An SAE was defined as any AE that was fatal, life threatening, requires prolonged inpatient hospitalization, resulted in significant disability or resulted in a congenital anomaly to a mother exposed to study treatment. AEs and SAEs were reported based on the NCI-CTCAE, v4.0. Percentages have been rounded off to the first decimal point.
Time Frame: From study start to 3 months after last dose of study drug (approximately 21 months)
Population: Safety-evaluable population included all participants who received at least one dose of any component of the combination. The safety-evaluable population in the DLBCL cohorts were assessed in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 3 | 6 | 8 | 40
percentage of participants
  AEs | 100 | 100 | 87.5 | 97.5
  SAEs | 100 | 66.7 | 25.0 | 30.0

4. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT=any one of the events that occurred in first treatment cycle & per the investigator was related to study treatment. Any AE that lead to a delay of > 14 days in start of next treatment cycle; Any Grade 3/4 non-hematologic AE with few exceptions; Any increase in hepatic transaminase >3×baseline(BL) & increase in direct bilirubin >2×upper limit of normal (ULN), without any findings of cholestasis/jaundice/signs of hepatic dysfunction & in absence of other contributory factors; Grade1 alanine transaminase (ALT)/aspartate transaminase (AST) elevation at BL as result of liver metastases, only a Grade ≥3 elevation, also ≥3×BL lasting >7 days; Hematologic AE meeting protocol specified criteria. Events were graded per NCI CTCAE v4.0. Grade 1:Mild; asymptomatic/mild symptoms; Grade 2:Moderate;minimal,local/non-invasive intervention indicated; Grade 3:Severe/medically significant, but not immediately life-threatening; Grade 4:Life-threatening consequences/urgent intervention indicated.
Time Frame: Day 1 of Cycle 1 to Day 1 of Cycle 2 (1 cycle=21 days) in dose-escalation phase
Population: Safety-evaluable population included all participants who received at least one dose of any component of the combination. The safety-evaluable population in the dose-escalation cohorts cohorts were assessed in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 3 | 6 | 8
Participants | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0

5. Primary Outcome: RP2D of Polatuzumab Vedotin
Description: RP2D was defined as the highest dose with acceptable toxicity as determined from dose-escalation phase. The RP2D of polatuzumab vedotin when given in combination with fixed dose of obinutuzumab in participants with FL was determined.
Time Frame: Day 1 of Cycle 1 to Day 1 of Cycle 2 (1 cycle=21 days) in dose-escalation phase
Population: as for outcome 2
Measure: Number; unit: mg/kg
Groups:
- All FL Participants: Dose Escalation: All participants with FL received venetoclax, at a dose of 200 mg, 400 mg, 600 mg or 800 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) in combination with obinutuzumab, 1000 mg, IV infusion, on Days 1, 8 and 15 of Cycle 1 and thereafter on Day 1 of Cycles 2-6 and polatuzumab vedotin, at a dose of 1.4 mg/kg or 1.8 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received venetoclax, at a dose of 200 mg, 400 mg, 600 mg or 800 mg, QD, for up to 8 months and obinutuzumab, 1000 mg on Day 1 of every other month (1 month=28 days) starting from Month 2 for up to 24 months.
Arm/Group | All FL Participants: Dose Escalation
Number analyzed (Participants) | 33
mg/kg | 1.8

6. Primary Outcome: RP2D of Venetoclax
Description: RP2D was defined as the highest dose with acceptable toxicity as determined from dose-escalation phase. The RP2D of venetoclax when given in combination with fixed dose of polatuzumab vedotin in participants with FL and DLBCL was determined.
Time Frame: Day 1 of Cycle 1 to Day 1 of Cycle 2 (1 cycle=21 days) in dose-escalation phase
Population: as for outcome 3
Measure: Number; unit: mg
Groups:
- All DLBCL Participants: Dose Escalation: All participants with DLBCL received venetoclax, at a dose of 400 mg, 600 mg or 800 mg, orally, QD on Days 1-21 of Cycles 1-6 (1 cycle=21 days) along with rituximab, 375 mg/m^2, IV infusion, on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, IV infusion, on Day 1 of Cycles 1-6 as induction treatment. Thereafter participants who achieved CR or PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 8 months. During consolidation treatment participants received venetoclax, at a dose of 400 mg, 600 mg or 800 mg, QD, for up to 8 months and rituximab, 375 mg/m^2 on Day 1 of every other month (1 month=28 days) starting from Month 2 up to 8 months.
Arm/Group | All FL Participants: Dose Escalation | All DLBCL Participants: Dose Escalation
Number analyzed (Participants) | 33 | 17
mg | 800 | 800

7. Secondary Outcome: Percentage of Participants With CR at EOI, Determined by the Investigator on the Basis of PET-CT Scans
Description: CR at EOI was assessed by Investigator according to MLRC. Per MLRC, CR based on PET-CT was defined as complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass, on 5PS where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake > mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions; no evidence of FDG-avid disease in bone marrow. 90% CI for percentage of responders was calculated using Clopper-Pearson method. Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 23 weeks) (1 cycle=21days)
Population: Efficacy evaluable population included participants in the dose expansion arms who received at least one dose of any component of the combination. As pre-specified in the protocol, participants who received polatuzumab vedotin and venetoclax at RP2D in dose-escalation phase were also analyzed in addition to expansion phase participants for efficacy analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 8 | 41 | 8 | 40
percentage of participants | 100 [68.77 to 100.00] | 51.2 [37.44 to 64.86] | 25.0 [4.64 to 59.97] | 32.5 [20.41 to 46.63]

8. Secondary Outcome: Percentage of Participants With CR at EOI, Determined by the IRC on the Basis of CT Scans Alone
Description: CR at EOI was determined by IRC according to the MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 centimeters (cm) in longest transverse diameter (LDi) and no ELS of disease; organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, immunohistochemistry (IHC) negative. 90% CI for percentage of responders was calculated using Clopper-Pearson method. Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 23 weeks) (1 cycle=21days)
Population: Efficacy evaluable population included participants in the dose expansion arms who received at least one dose of any component of the combination. As pre-specified in the protocol, participants who received polatuzumab vedotin and venetoclax at RP2D in dose-escalation phase were also analyzed in addition to expansion phase participants for efficacy analysis. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 8 | 41 | 6 | 34
percentage of participants | 62.5 [28.92 to 88.89] | 36.6 [24.08 to 50.61] | 16.7 [0.85 to 58.18] | 26.5 [14.56 to 41.65]

9. Secondary Outcome: Percentage of Participants With CR at EOI, Determined by the Investigator on the Basis of CT Scans Alone
Description: CR at EOI was determined by Investigator according to the MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease; organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. 90% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 23 weeks) (1 cycle=21days)
Population: as for outcome 7
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 8 | 41 | 8 | 40
percentage of participants | 75.0 [40.03 to 95.36] | 29.3 [17.84 to 43.07] | 25.0 [4.64 to 59.97] | 22.5 [12.27 to 35.98]

10. Secondary Outcome: Percentage of Participants With Objective Response (OR) at EOI, Determined by an IRC on the Basis of PET and CT Scans
Description: OR=percentage of participants with CR or PR as assessed by the IRC according to MLRC. Per MLRC CR based on PET-CT=complete MR in lymph nodes & ELS with score of 1, 2, or 3 with or without residual mass on 5PS, where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake> mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions; no new lesions & no evidence of FDG-avid disease in bone marrow. PR based on PET-CT=partial MR in lymph nodes & ELS with score of 4 or 5 with reduced uptake compared with baseline & residual masses of any size: at interim (suggest responding disease) or at end of treatment (indicate residual disease), residual uptake higher than uptake in normal bone marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed). 90% CI was calculated using Clopper-Pearson method. Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 23 weeks) (1 cycle=21days)
Population: as for outcome 7
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 8 | 41 | 8 | 40
percentage of participants | 100.0 [68.77 to 100.00] | 70.7 [56.93 to 82.16] | 25.0 [4.64 to 59.97] | 37.5 [24.73 to 51.72]

11. Secondary Outcome: Percentage of Participants With OR at EOI, Determined by the Investigator on the Basis of PET and CT Scans
Description: OR=percentage of participants with CR or PR as assessed by the IRC according to MLRC. Per MLRC CR based on PET-CT=complete MR in lymph nodes & ELS with score of 1, 2, or 3 with or without residual mass on 5PS, where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake> mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions;no new lesions & no evidence of FDG-avid disease in bone marrow. PR based on PET-CT=partial MR in lymph nodes & ELS with score of 4 or 5 with reduced uptake compared with baseline & residual masses of any size: at interim (suggest responding disease) or at end of treatment (indicate residual disease), residual uptake higher than uptake in normal bone marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed). 90% CI was calculated using Clopper-Pearson method. Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 23 weeks) (1 cycle=21days)
Population: as for outcome 7
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 8 | 41 | 8 | 40
percentage of participants | 100.0 [68.77 to 100.00] | 75.6 [62.15 to 86.13] | 37.5 [11.11 to 71.08] | 42.5 [29.18 to 56.69]

12. Secondary Outcome: Percentage of Participants With OR at EOI, Determined by an IRC on the Basis of CT Scans Alone
Description: OR was defined as the percentage of participants with CR or PR, as assessed by the IRC based on MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease; organ enlargement regressing to normal; no new lesions; bone marrow normal by morphology, if indeterminate, IHC negative. PR per CT only was defined as partial remission in lymph nodes and ELS with ≥50% decrease in the sum of the products of greatest diameters (SPD) of up to 6 target measurable lymph nodes and extranodal sites, absent/normal/regressed but with no increase in non-measured lesions, spleen regressing by ≥50% in length beyond normal, no new sites of lesions. 90% CI for percentage of responders was calculated using Clopper-Pearson method. Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 23 weeks) (1 cycle=21days)
Population: as for outcome 7
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 8 | 41 | 8 | 40
percentage of participants | 87.5 [52.93 to 99.36] | 82.9 [70.31 to 91.70] | 25.0 [4.64 to 59.97] | 37.5 [24.73 to 51.72]

13. Secondary Outcome: Percentage of Participants With OR at EOI, Determined by the Investigator on the Basis of CT Scans Alone
Description: OR was defined as the percentage of participants with CR or PR, as assessed by the investigator based on MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease; organ enlargement regressing to normal; no new lesions; bone marrow normal by morphology, if indeterminate, IHC negative. PR per CT only was defined as partial remission in lymph nodes and ELS with ≥50% decrease in the SPD of up to 6 target measurable lymph nodes and extranodal sites, absent/normal/regressed but with no increase in non-measured lesions, spleen regressing by ≥50% in length beyond normal, no new sites of lesions. 90% CI for percentage of responders was calculated using Clopper-Pearson method. Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 23 weeks) (1 cycle=21days)
Population: as for outcome 7
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 8 | 41 | 8 | 40
percentage of participants | 87.5 [52.93 to 99.36] | 85.4 [73.15 to 93.43] | 37.5 [11.11 to 71.08] | 45.0 [31.46 to 59.12]

14. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) of CR or PR, Determined by the Investigator on the Basis of CT Scans Alone
Description: BOR=CR or PR as assessed by investigator per CT per MLRC. Per MLRC, CR based on CT was defined as a complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease; organ enlargement regressing to normal; no new lesions; bone marrow normal by morphology, if indeterminate, IHC negative. PR per CT only was defined as partial remission in lymph nodes and ELS with ≥50% decrease in SPD of up to 6 target measurable lymph nodes and extranodal sites, absent/normal/regressed but with no increase in non-measured lesions, spleen regressing by ≥50% in length beyond normal, no new sites of lesions. Percentages have been rounded off to the first decimal point.
Time Frame: Up to every 6 months until disease progression, the start of new anti-lymphoma treatment, or the end of the study, whichever occurs first (approximately 77 months)
Population: as for outcome 7
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 8 | 41 | 8 | 40
percentage of participants | 100.0 [68.77 to 100.00] | 87.8 [76.05 to 95.07] | 50.0 [19.29 to 80.71] | 72.5 [58.61 to 83.75]

15. Secondary Outcome: Observed Serum Obinutuzumab Concentration
Time Frame: Pre-dose & 0.5 hours post-dose on Day 1 Cycles 1, 2, 4, & 6; and pre-dose on Day 1 of Months 2, 8, 14, 20; study drug discontinuation, Day 120 &1 year post-last dose (up to approximately 40 months) (1 cycle = 21 days)
Population: Pharmacokinetics (PK) evaluable population included all participants who had at least one evaluable PK sample post dose for at least one analyte. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 39
micrograms per milliliter (µg/mL)
  Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 6 | 3 | 3 | 3 | 9 | 8 | 29
  Cycle 1 Day 1: Pre-dose | NA (NA) — The data was not evaluable as the samples were below lower limit of quantification (BLLQ). | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ.
  Cycle 1 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 5 | 3 | 3 | 3 | 9 | 5 | 38
  Cycle 1 Day 1: 0.5 hours Post Dose | 310 (21.2) | 360 (18.8) | 169 (60.2) | 342 (11.0) | 262 (106.0) | 438 (17.8) | 261 (115.1)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 39
  Cycle 2 Day 1: Pre-dose | 327 (46.7) | 498 (20.6) | 288 (43.2) | 395 (17.0) | 435 (25.4) | 497 (20.3) | 422 (29.0)
  Cycle 2 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 39
  Cycle 2 Day 1: 0.5 hours Post Dose | 637 (32.0) | 822 (17.0) | 512 (56.1) | 685 (17.8) | 800 (19.1) | 975 (19.3) | 834 (30.3)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 7 | 36
  Cycle 4 Day 1: Pre-dose | 284 (50.9) | 496 (25.3) | 376 (9.6) | 337 (12.0) | 422 (20.3) | 454 (37.2) | 397 (40.5)
  Cycle 4 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 7 | 36
  Cycle 4 Day 1: 0.5 hours Post Dose | 534 (62.9) | 842 (25.1) | 709 (20.1) | 732 (13.4) | 819 (18.6) | 925 (26.9) | 770 (25.6)
  Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 7 | 36
  Cycle 6 Day 1: Pre-dose | 288 (62.9) | 582 (26.5) | 338 (4.0) | 335 (10.2) | 437 (24.5) | 420 (44.5) | 428 (51.9)
  Cycle 6 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 6 | 3 | 2 | 3 | 8 | 7 | 36
  Cycle 6 Day 1: 0.5 hours Post Dose | 582 (26.8) | 887 (19.6) | 490 (65.2) | 659 (14.3) | 857 (21.2) | 841 (28.1) | 807 (27.0)
  Maintenance Month 2: number analyzed (Participants) | 6 | 3 | 1 | 3 | 8 | 7 | 31
  Maintenance Month 2 | 117 (471.2) | 294 (53.3) | 205 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 192 (11.7) | 273 (63.4) | 327 (57.6) | 291 (60.8)
  Maintenance Month 8: number analyzed (Participants) | 3 | 1 | 1 | 2 | 7 | 6 | 20
  Maintenance Month 8 | 148 (161.8) | 184 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 191 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 114 (30.0) | 170 (40.2) | 210 (27.0) | 168 (72.0)
  Maintenance Month 14: number analyzed (Participants) | 2 | 2 | 1 | 1 | 4 | 2 | 14
  Maintenance Month 14 | 189 (112.9) | 226 (28.9) | 197 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 138 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 133 (23.5) | 190 (17.9) | 168 (41.3)
  Maintenance Month 20: number analyzed (Participants) | 1 | 2 | 1 | 0 | 4 | 4 | 12
  Maintenance Month 20 | 242 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 218 (30.7) | 74.0 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |  | 156 (44.2) | 144 (26.9) | 180 (62.0)
  Study Drug Discontinuation Visit: number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 4 | 16
  Study Drug Discontinuation Visit | 9.61 (438943.9) | 134 (1414.6) | 4.48 (2973890.2) | 66.6 (271.0) | 262 (11.9) | 212 (34.8) | 148 (110.1)
  Day 120 Post Last Dose: number analyzed (Participants) | 1 | 0 | 3 | 1 | 4 | 5 | 10
  Day 120 Post Last Dose | 39.9 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |  | 1.72 (1634893.3) | 0.660 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 41.2 (89.5) | 94.6 (85.6) | 44.1 (274.2)
  One Year Post Last Dose: number analyzed (Participants) | 4 | 0 | 2 | 1 | 3 | 1 | 6
  One Year Post Last Dose | 0.0410 (20351.2) |  | 0.0585 (372.7) | 0.00680 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.244 (716.1) | 0.0820 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 4.89 (9002.8)

16. Secondary Outcome: Observed Serum Rituximab Concentration
Time Frame: Pre-dose and 0.5 hours post-dose on Day 1 of Cycles 1 and 6; pre-dose on Day 1 of Cycles 2 and 4; (1 cycle = 21 days)
Population: PK-evaluable population included all participants who had at least one evaluable PK sample post dose for at least one analyte. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 2 | 6 | 6 | 39
µg/mL
  Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 2 | 2 | 1 | 9
  Cycle 1 Day 1: Pre-dose | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ.
  Cycle 1 Day 1: 0.5 hours Post Dose | 199 (25.4) | 189 (6.8) | 255 (14.0) | 146 (159.3)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 2 | 6 | 6 | 36
  Cycle 2 Day 1: Pre-dose | 49.3 (17.2) | 38.9 (61.7) | 71.0 (42.1) | 50.1 (30.5)
  Cycle 4 Day 1:Pre-dose: number analyzed (Participants) | 2 | 2 | 4 | 29
  Cycle 4 Day 1:Pre-dose | 88.9 (11.1) | 39.3 (71.0) | 126 (16.5) | 88.1 (43.4)
  Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 2 | 1 | 3 | 24
  Cycle 6 Day 1: Pre-dose | 120 (8.8) | 20.9 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 151 (32.4) | 117 (43.4)
  Cycle 6 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 2 | 1 | 3 | 23
  Cycle 6 Day 1: 0.5 hours Post Dose | 303 (12.4) | 182 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 229 (36.9) | 308 (27.2)

17. Secondary Outcome: Observed Serum Concentration of Total Antibody to Polatuzumab Vedotin
Description: Total antibody is an analyte of polatuzumab vedotin.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2 and 4; study drug discontinuation visit; Day 120 and 1 year post-last dose (up to approximately 16 months) (1 cycle=21 days)
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 41 | 3 | 6 | 7 | 39
µg/mL
  Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 7 | 41 | 2 | 6 | 7 | 39
  Cycle 1 Day 1: Pre-dose | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ.
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 40 | 3 | 6 | 6 | 37
  Cycle 2 Day 1: Pre-dose | 0.798 (404.2) | 3.14 (29.4) | 0.677 (6220.9) | 2.03 (46.4) | 1.75 (63.2) | 4.22 (31.1) | 1.73 (265.3) | 3.34 (56.6) | 2.23 (83.5) | 3.41 (30.9) | 3.04 (70.8)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 7 | 36 | 3 | 2 | 4 | 30
  Cycle 4 Day 1: Pre-dose | 2.73 (76.1) | 6.12 (26.1) | 7.88 (9.5) | 5.40 (18.4) | 5.72 (33.5) | 8.19 (32.3) | 5.88 (63.7) | 6.84 (29.5) | 2.34 (82.1) | 8.22 (17.0) | 5.82 (45.7)
  Study Drug Discontinuation Visit: number analyzed (Participants) | 2 | 2 | 2 | 3 | 4 | 4 | 17 | 1 | 1 | 4 | 14
  Study Drug Discontinuation Visit | 0.0250 (NA) — Values were less than reportable (LTR) for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 0.0250 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 0.0534 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 0.0250 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0250 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0900 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.110 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 2.43 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 4.71 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 1.38 (203.0) | 1.03 (471.1)
  Day 120 Post Last Dose: number analyzed (Participants) | 1 | 1 | 3 | 1 | 6 | 6 | 20 | 2 | 0 | 1 | 7
  Day 120 Post Last Dose | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.0906 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.0832 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.156 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.494 (468.8) | 0.385 (28.6) |  | 0.759 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 1.37 (93.2)
  One Year Post Last Dose: number analyzed (Participants) | 4 | 0 | 2 | 1 | 3 | 1 | 11 | 1 | 1 | 0 | 3
  One Year Post Last Dose | 0.0250 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. |  | 0.0250 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.0250 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.0294 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |  | 0.0457 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable.

18. Secondary Outcome: Observed Plasma Concentration of Polatuzumab Vedotin Antibody-Conjugated Mono-Methyl Auristatin E (MMAE) (acMMAE)
Description: acMMAE is an analyte of polatuzumab vedotin.
Time Frame: Pre-dose and 0.5 hours post-dose on Day 1 of Cycles 1, 2 and 4; post-dose on Days 8 and 15 of Cycle 1; predose on Day 1 of Cycle 6 (1 cycle=21 days)
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 40 | 3 | 6 | 8 | 39
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1: Pre-dose | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Cycle 1 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 6 | 3 | 3 | 3 | 9 | 8 | 39 | 3 | 6 | 8 | 38
  Cycle 1 Day 1: 0.5 hours Post Dose | 131 (19054.2) | 530 (22.2) | 451 (48.0) | 610 (3.4) | 645 (24.6) | 825 (20.8) | 613 (38.2) | 722 (25.3) | 628 (27.1) | 683 (22.2) | 481 (226.7)
  Cycle 1 Day 8: Post Dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 40 | 2 | 5 | 6 | 36
  Cycle 1 Day 8: Post Dose | 19.1 (890.8) | 57.0 (19.3) | 9.87 (43972.4) | 49.3 (33.6) | 58.0 (39.7) | 88.9 (20.7) | 41.0 (192.1) | 45.6 (27.7) | 50.8 (42.6) | 77.0 (25.3) | 57.9 (42.2)
  Cycle 1 Day 15: Post Dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 39 | 3 | 6 | 6 | 37
  Cycle 1 Day 15: Post Dose | 6.67 (421.2) | 22.9 (18.1) | 4.56 (5235.8) | 18.7 (24.2) | 17.7 (56.9) | 31.6 (15.3) | 14.4 (176.9) | 26.0 (69.8) | 19.8 (50.5) | 30.2 (21.5) | 22.3 (40.6)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 39 | 3 | 5 | 6 | 35
  Cycle 2 Day 1: Pre-dose | 3.69 (296.8) | 12.6 (36.9) | 3.25 (2446.9) | 9.34 (44.7) | 8.27 (62.6) | 16.7 (40.2) | 7.71 (209.4) | 14.9 (66.9) | 8.94 (100.6) | 14.8 (29.2) | 13.1 (45.3)
  Cycle 2 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 39 | 3 | 6 | 6 | 37
  Cycle 2 Day 1: 0.5 hours Post Dose | 527 (27.3) | 594 (18.7) | 602 (36.8) | 555 (3.0) | 682 (24.0) | 844 (19.7) | 688 (20.7) | 749 (23.0) | 341 (353.1) | 748 (17.7) | 628 (27.6)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 7 | 37 | 3 | 2 | 4 | 30
  Cycle 4 Day 1: Pre-dose | 10.8 (69.4) | 18.8 (24.9) | 29.4 (10.1) | 19.7 (8.2) | 23.4 (35.0) | 27.5 (37.0) | 21.5 (53.3) | 24.8 (25.8) | 8.16 (245.5) | 30.1 (12.3) | 22.2 (49.8)
  Cycle 4 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 6 | 37 | 3 | 2 | 4 | 29
  Cycle 4 Day 1: 0.5 hours Post Dose | 491 (28.1) | 587 (16.3) | 768 (29.5) | 620 (7.4) | 553 (90.9) | 474 (299.3) | 644 (66.8) | 968 (33.7) | 722 (1.8) | 775 (15.2) | 680 (25.9)
  Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 7 | 33 | 2 | 1 | 3 | 24
  Cycle 6 Day 1: Pre-dose | 13.0 (58.5) | 4.62 (5273.1) | 23.5 (42.5) | 20.5 (3.7) | 28.6 (27.2) | 27.3 (35.9) | 25.2 (56.9) | 24.3 (24.4) | 3.73 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 31.5 (46.0) | 24.7 (54.4)

19. Secondary Outcome: Observed Plasma Concentration of Polatuzumab Vedotin Unconjugated MMAE
Description: MMAE is an analyte of polatuzumab vedotin.
Time Frame: as for outcome 18
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 40 | 3 | 6 | 8 | 38
ng/mL
  Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 39 | 3 | 6 | 8 | 38
  Cycle 1 Day 1: Pre-dose | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ. | NA (NA) — The data was not evaluable as the samples were BLLQ.
  Cycle 1 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 6 | 3 | 3 | 3 | 9 | 8 | 40 | 3 | 6 | 8 | 38
  Cycle 1 Day 1: 0.5 hours Post Dose | 0.313 (725.2) | 0.236 (31.1) | 1.04 (575.7) | 0.417 (60.3) | 0.507 (112.0) | NA (NA) — The data was not evaluable as the samples were BLLQ | 0.441 (208.3) | 0.249 (8.7) | 0.390 (89.0) | 0.262 (61.9) | 0.263 (90.8)
  Cycle 1 Day 8: Post Dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 40 | 3 | 5 | 6 | 36
  Cycle 1 Day 8: Post Dose | 1.14 (34.8) | 57.5 (1.46) | 1.57 (63.6) | 1.06 (43.6) | 1.66 (69.9) | 0.323 (79.3) | 1.81 (65.3) | 2.34 (54.7) | 2.77 (63.1) | 2.51 (96.3) | 2.51 (65.1)
  Cycle 1 Day 15: Post Dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 39 | 3 | 6 | 6 | 37
  Cycle 1 Day 15: Post Dose | 0.225 (87.4) | 0.310 (60.2) | 0.213 (174.3) | 0.341 (55.9) | 0.461 (76.6) | 2.26 (76.3) | 0.444 (99.8) | 0.675 (144.7) | 0.927 (89.8) | 0.778 (77.9) | 0.723 (63.3)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 39 | 3 | 6 | 6 | 37
  Cycle 2 Day 1: Pre-dose | 0.0575 (117.0) | 0.103 (47.1) | 0.0565 (132.5) | 0.0982 (75.3) | 0.0866 (141.8) | 0.688 (73.8) | 0.113 (136.1) | 0.221 (199.1) | 0.311 (76.4) | 0.266 (161.7) | 0.227 (66.1)
  Cycle 2 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 39 | 3 | 6 | 6 | 37
  Cycle 2 Day 1: 0.5 hours Post Dose | 0.152 (46.2) | 0.184 (29.0) | 0.399 (104.7) | 0.175 (57.0) | 0.231 (76.5) | 0.150 (41.9) | 0.257 (63.8) | 0.343 (122.0) | 0.564 (76.4) | 0.407 (116.2) | 0.322 (55.9)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 8 | 36 | 3 | 2 | 4 | 30
  Cycle 4 Day 1: Pre-dose | 0.131 (58.2) | 0.106 (48.3) | 0.180 (62.4) | 0.172 (46.8) | 0.155 (46.5) | 0.263 (46.5) | 0.167 (81.0) | 0.238 (75.5) | 0.459 (103.4) | 0.295 (90.5) | 0.220 (72.7)
  Cycle 4 Day 1: 0.5 hours Post Dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 7 | 37 | 3 | 2 | 4 | 29
  Cycle 4 Day 1: 0.5 hours Post Dose | 0.235 (84.2) | 0.163 (50.6) | 0.255 (48.6) | 0.270 (31.6) | 0.209 (42.0) | 0.206 (36.2) | 0.260 (56.2) | 0.331 (77.4) | 0.565 (107.5) | 0.364 (65.6) | 0.311 (57.7)
  Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 6 | 35 | 2 | 1 | 2 | 24
  Cycle 6 Day 1: Pre-dose | 0.107 (73.4) | 0.120 (62.3) | 0.0715 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 0.239 (17.2) | 0.189 (37.2) | 0.289 (55.2) | 0.162 (94.9) | 0.197 (275.2) | 0.795 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.334 (62.1) | 0.211 (93.8)

20. Secondary Outcome: Observed Plasma Venetoclax Concentration
Time Frame: Pre-dose and 4 hours post-dose on Day 1 Cycle 1, pre-dose & 2, 4, 6, & 8 hours post-dose on Day 1 Cycle 2, pre-dose & 4hours post-dose on Day 1 Cycle 4 & pre-dose on Day 1 Cycle 6; (1 cycle = 21 days)
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 41 | 3 | 6 | 7 | 40
µg/mL
  Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Cycle 1 Day 1: Pre-dose |  |  |  |  |  |  |  |  |  |  | NA (NA) — The data was not evaluable as the samples were BLLQ.
  Cycle 1 Day 1: Post Dose: number analyzed (Participants) | 6 | 3 | 3 | 3 | 9 | 8 | 41 | 3 | 6 | 7 | 40
  Cycle 1 Day 1: Post Dose | 0.624 (94.6) | 0.247 (162.1) | 0.108 (53.3) | 0.244 (149.1) | 0.796 (86.5) | 0.811 (310.3) | 0.964 (69.2) | 0.503 (47.9) | 0.915 (47.4) | 1.21 (103.4) | 0.841 (94.8)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 39 | 3 | 6 | 6 | 35
  Cycle 2 Day 1: Pre-dose | 0.336 (99.3) | 0.347 (144.3) | 0.453 (71.9) | 0.943 (28.5) | 0.298 (2853.1) | 0.282 (498.3) | 0.555 (1134.4) | 0.529 (135.6) | 0.952 (139.7) | 0.852 (1812.3) | 0.329 (1047.7)
  Cycle 2 Day 1: 2 hours Post Dose: number analyzed (Participants) | 7 | 3 | 2 | 2 | 7 | 6 | 1 | 3 | 5 | 5 | 1
  Cycle 2 Day 1: 2 hours Post Dose | 0.532 (119.2) | 0.306 (107.3) | 0.351 (129.3) | 0.822 (54.8) | 0.769 (131.0) | 0.921 (74.0) | 2.69 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.632 (90.1) | 1.08 (82.0) | 1.01 (464.7) | NA (5.13) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.
  Cycle 2 Day 1: 4 hours Post Dose: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 7 | 39 | 3 | 6 | 6 | 37
  Cycle 2 Day 1: 4 hours Post Dose | 1.12 (102.2) | 0.572 (49.1) | 0.548 (51.0) | 1.31 (22.5) | 1.65 (69.4) | 2.04 (39.2) | 1.99 (59.0) | 0.830 (75.3) | 1.49 (43.1) | 2.03 (131.4) | 1.50 (74.5)
  Cycle 2 Day 1: 6 hours Post Dose: number analyzed (Participants) | 7 | 3 | 2 | 2 | 7 | 6 | 1 | 3 | 5 | 5 | 1
  Cycle 2 Day 1: 6 hours Post Dose | 1.38 (83.4) | 0.933 (72.1) | 1.21 (24.8) | 1.99 (5.7) | 2.15 (51.9) | 2.55 (28.0) | 4.82 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.870 (98.1) | 1.96 (57.5) | 2.74 (117.9) | 5.95 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.
  Cycle 2 Day 1: 8 hours Post Dose: number analyzed (Participants) | 7 | 3 | 2 | 2 | 6 | 5 | 1 | 3 | 4 | 4 | 1
  Cycle 2 Day 1: 8 hours Post Dose | 1.40 (74.9) | 0.803 (76.7) | 1.45 (32.3) | 2.24 (18.4) | 2.46 (59.8) | 2.53 (32.7) | 3.02 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.886 (87.6) | 1.88 (70.8) | 2.85 (94.7) | 6.66 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 7 | 36 | 3 | 2 | 4 | 30
  Cycle 4 Day 1: Pre-dose | 0.259 (157.2) | 0.0344 (15072.4) | 0.302 (1.2) | 1.12 (40.2) | 0.551 (98.4) | 0.304 (1059.7) | 0.561 (401.2) | 0.0581 (1105.7) | 0.933 (74.2) | 0.826 (311.3) | 0.337 (1043.6)
  Cycle 4 Day 1: Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Cycle 4 Day 1: Post Dose |  |  |  |  |  |  |  |  |  |  | 1.04 (8.4)
  Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 7 | 3 | 2 | 3 | 8 | 7 | 34 | 2 | 1 | 3 | 24
  Cycle 6 Day 1: Pre-dose | 0.252 (95.0) | 0.277 (178.7) | 0.0177 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 1.24 (56.1) | 0.595 (95.4) | 0.0266 (26843.8) | 0.509 (496.6) | 0.175 (187.9) | 1.90 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.0772 (101668.3) | 0.365 (780.9)

21. Secondary Outcome: Number of Participants With Human Anti-Human Antibodies (HAHAs) to Obinutuzumab
Description: The number of participants with positive results for HAHAs, also called anti-drug antibodies (ADAs) against obinutuzumab at baseline and at any of the post-baseline assessment time-points were reported. Number of participants positive for Treatment Emergent ADA = the number of post-baseline evaluable participants determined to have treatment induced ADA or treatment-enhanced ADA during the study period. Treatment-induced ADA = negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at baseline who has one or more post-baseline titer results that are at least 0.60 titer unit (t.u.) greater than the baseline titer result.
Time Frame: Baseline up to approximately 2 years after last dose (up to approximately 56 months)
Population: The immunogenicity population included participants with at least one predose and one postdose HAHA or ATA assessment, with participants grouped according to histology. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 39
Participants
  Baseline prevalence of ADAs: number analyzed (Participants) | 7 | 3 | 2 | 3 | 9 | 7 | 39
  Baseline prevalence of ADAs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post baseline incidence of ADAs: number analyzed (Participants) | 7 | 3 | 3 | 3 | 8 | 8 | 39
  Post baseline incidence of ADAs | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Anti-Therapeutic Antibodies (ATAs) to Polatuzumab Vedotin
Description: The number of participants with positive results for ATAs, also called ADAs against polatuzumab vedotin at baseline and at any of the post-baseline assessment time-points were reported. Number of participants positive for Treatment Emergent ADA = the number of post-baseline evaluable participants determined to have treatment induced ADA or treatment-enhanced ADA during the study period. Treatment-induced ADA = negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at baseline who has one or more post-baseline titer results that are at least 0.60 t.u. greater than the baseline titer result.
Time Frame: Baseline up to 1 year post last dose (up to approximately 16 months)
Population: Immunogenicity population included participants with at least one predose and one postdose HAHA or ATA assessment, with participants grouped according to histology. Number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
Number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 41 | 3 | 6 | 8 | 40
Participants
  Baseline prevalence of ADAs: number analyzed (Participants) | 6 | 3 | 3 | 3 | 9 | 7 | 41 | 3 | 6 | 8 | 40
  Baseline prevalence of ADAs | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post baseline incidence of ADAs: number analyzed (Participants) | 7 | 3 | 3 | 3 | 9 | 8 | 41 | 3 | 6 | 7 | 39
  Post baseline incidence of ADAs | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: FL cohorts: From study start to 24 months after last dose of study drug (approximately 56 months); DLBCL cohorts: From study start to 3 months after last dose of study drug (approximately 21 months)
Description: Safety-evaluable population included all participants who received at least one dose of any component of the combination.
Arm/Group | FL Dose Escalation: 1.4P+400V+1000G | FL Dose Escalation: 1.4P+200V+1000G | FL Dose Escalation: 1.8P+400V+1000G | FL Dose Escalation: 1.4P+600V+1000G | FL Dose Escalation: 1.8P+600V+1000G | FL Dose Escalation: 1.8P+800V+1000G | FL: Dose Expansion: 1.8P+800V+1000G | DLBCL: Dose Escalation: 1.8P+400V+375R | DLBCL Dose Escalation: 1.8P+600V+375R | DLBCL Dose Escalation: 1.8P+800V+375R | DLBCL Dose Expansion: 1.8P+800V+375R
All-Cause Mortality (participants affected / at risk) | 3/7 | 1/3 | 0/3 | 0/3 | 1/9 | 1/8 | 8/41 | 0/3 | 4/6 | 6/8 | 26/40
Serious Adverse Events (participants affected / at risk) | 4/7 | 1/3 | 1/3 | 0/3 | 2/9 | 6/8 | 14/41 | 3/3 | 4/6 | 2/8 | 12/40
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 3/3 | 3/3 | 9/9 | 8/8 | 41/41 | 3/3 | 6/6 | 7/8 | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FL Dose Escalation: 1.4P+400V+1000G (N=7) | FL Dose Escalation: 1.4P+200V+1000G (N=3) | FL Dose Escalation: 1.8P+400V+1000G (N=3) | FL Dose Escalation: 1.4P+600V+1000G (N=3) | FL Dose Escalation: 1.8P+600V+1000G (N=9) | FL Dose Escalation: 1.8P+800V+1000G (N=8) | FL: Dose Expansion: 1.8P+800V+1000G (N=41) | DLBCL: Dose Escalation: 1.8P+400V+375R (N=3) | DLBCL Dose Escalation: 1.8P+600V+375R (N=6) | DLBCL Dose Escalation: 1.8P+800V+375R (N=8) | DLBCL Dose Expansion: 1.8P+800V+375R (N=40)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL TEAR (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADVERSE DRUG REACTION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE LEAKAGE (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FL Dose Escalation: 1.4P+400V+1000G (N=7) | FL Dose Escalation: 1.4P+200V+1000G (N=3) | FL Dose Escalation: 1.8P+400V+1000G (N=3) | FL Dose Escalation: 1.4P+600V+1000G (N=3) | FL Dose Escalation: 1.8P+600V+1000G (N=9) | FL Dose Escalation: 1.8P+800V+1000G (N=8) | FL: Dose Expansion: 1.8P+800V+1000G (N=41) | DLBCL: Dose Escalation: 1.8P+400V+375R (N=3) | DLBCL Dose Escalation: 1.8P+600V+375R (N=6) | DLBCL Dose Escalation: 1.8P+800V+375R (N=8) | DLBCL Dose Expansion: 1.8P+800V+375R (N=40)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 7 (13) | 1 (1) | 2 (3) | 3 (4) | 5 (9)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGAMMAGLOBULINAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (9)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (3) | 1 (3) | 2 (2) | 1 (5) | 4 (17) | 5 (23) | 17 (46) | 2 (5) | 2 (7) | 5 (7) | 20 (64)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (8) | 12 (37) | 1 (1) | 0 (0) | 1 (1) | 6 (8)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
DEAFNESS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTORRHOEA (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIPLOPIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCLERAL HYPERAEMIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (6) | 0 (0) | 1 (2) | 3 (3) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 10 (14) | 0 (0) | 2 (2) | 1 (2) | 6 (6)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (6) | 2 (2) | 3 (7) | 2 (2) | 5 (8) | 6 (14) | 20 (42) | 3 (4) | 1 (1) | 5 (8) | 16 (20)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FAECES SOFT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MUCOUS STOOLS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 4 (6) | 23 (35) | 3 (4) | 3 (4) | 1 (1) | 14 (15)
ODYNOPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL DISCHARGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2) | 2 (3) | 1 (2) | 3 (4) | 11 (17) | 2 (3) | 3 (3) | 4 (11) | 8 (8)
ADVERSE DRUG REACTION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
CHILLS (General disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
EARLY SATIETY (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 5 (7) | 2 (2) | 2 (2) | 1 (2) | 2 (2) | 3 (3) | 13 (14) | 1 (1) | 1 (1) | 3 (3) | 10 (10)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE BRUISING (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE EXTRAVASATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OEDEMA MUCOSAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (7) | 5 (5) | 1 (1) | 2 (3) | 2 (2) | 6 (7)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERIAL DISEASE CARRIER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CAMPYLOBACTER INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
CHRONIC SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 4 (6) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (3) | 11 (18) | 0 (0) | 1 (1) | 3 (4) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 4 (4) | 1 (1) | 13 (14) | 1 (2) | 0 (0) | 3 (4) | 2 (2)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN WOUND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUNBURN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VASCULAR ACCESS SITE PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AMYLASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BILIRUBIN CONJUGATED INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CALCIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CALCIUM INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
BLOOD FIBRINOGEN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BLOOD IMMUNOGLOBULIN G DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OCCULT BLOOD POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROTEIN TOTAL DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROTEIN URINE PRESENT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RED BLOOD CELLS URINE POSITIVE (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY CASTS PRESENT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (6) | 1 (1) | 3 (3) | 4 (5) | 6 (7)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
GOUT (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 4 (5) | 0 (0) | 4 (4) | 3 (3) | 4 (5)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 4 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 3 (8) | 7 (8) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 4 (8) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OCULAR MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OCULAR SURFACE SQUAMOUS NEOPLASIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (5) | 8 (15) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 3 (3) | 11 (11) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
PARAESTHESIA (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 1 (2) | 0 (0) | 3 (4)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESTING TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
TASTE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
INSOMNIA (Psychiatric disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (7) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
LIBIDO DECREASED (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
URINARY TRACT PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINE ABNORMALITY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANISOMASTIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CYST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENDOMETRIAL THICKENING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATIC DISORDER (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 1 (1) | 1 (3) | 1 (1) | 3 (3) | 4 (7) | 11 (14) | 2 (2) | 1 (1) | 0 (0) | 9 (11)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MILIARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 4 (7) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN HYPERTROPHY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SOLAR LENTIGO (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH EXTRACTION (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
POOR VENOUS ACCESS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUPERFICIAL VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT02611323/Prot_SAP_000.pdf